CLINICAL TRIAL: NCT04916457
Title: Explore the Role of Skin Microecology in Diabetic Skin Lesions Based on Multi-omics Data Analysis
Brief Title: The Role of Skin Microecology in Diabetic Skin Lesions
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-306
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot; Diabetic Dermopathy
Keywords: Diabetic foot; skin micro-ecology
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skin cotton sample, skin tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- group ND: control group without DM non-intervention
- group VD: very low-risk group: diabetic patient with no loss of protective sensation(LOPS) and no peripheral artery disease(PAD).
  non-intervention
- group LD: low-risk group: diabetic patient with LOPS or PAD non-intervention
- group MD: moderate-risk group: diabetic patient with LOPS + PAD non-intervention
- group HD: high-risk group: diabetic patient with LOPS or PAD, and one or more of the following:
  * history of a foot ulcer
  * a lower-extremity amputation (minor or major)
  * end-stage renal disease
  non-intervention

SUMMARY:
This study is an observational study. Collect cotton swabs of the surface skin are obtained from the non-diabetic and diabetic patients hospitalized in the Nanfang Hospital of Southern Medical University. The investigators use omics technology to identify the structure and functions of cutaneous microbiome, analyze the characteristics of the skin flora of diabetic patients, and find the difference in skin microbiota among diabetic patients with different risk levels for developing into diabetic foot. Then, the participants will be followed up to compare the incidence of ulcers among different groups. And the skin tissues discarded during surgical operations of non-diabetic and diabetes patients are collected for pathological examination. Finally, based on the results of 16S high-throughput sequencing, metagenomics, etc., specific flora could be extracted from human skin flora cotton swabs, and animal experiments are performed to explore the effect of skin micro-ecology on diabetic skin lesions. The investigators will explore in animal experiments to regulate the influence of skin micro-ecology on diabetic skin lesions through treatment methods such as different hypoglycemic drugs and probiotic emulsions.

DETAILED DESCRIPTION:
The study intends to explore the mechanism of diabetic skin micro-ecology in diabetic skin diseases, and find new ways of early screening and prevention for diabetic foot.

This study is a prospective observational study. Adult participants were divided into the following 5 groups (n=200, 40 in each group): control group, very low-risk group, low-risk group, moderate-risk group, and high-risk group. Sterile rayon tipped swabs were pre-moistened with a sterile solution containing 0.15 M NaCl and 0.1% Tween 20. All swabs samples were collected from the intact skin at plantar anterior. And the skin cotton swab was subjected to 16s rDNA high-throughput sequencing, metagenomic sequencing methods, etc. Based on the result, the investigators will analyse the change of the cutaneous microbiome in DM as the disease condition progresses.

The skin tissues of the control group and observation group who met the inclusion criteria were also collected during surgical operations, and pathological and immunohistochemistry tests were performed respectively to analyze the pathological changes of diabetic skin tissues in different disease progressions.

According to the results of multi-omics analysis, the research team screen for the specific flora. Then sort out and culture specific strains, and establish mouse model of microbiota transplantation in order to explore the effects of regulating skin microecology on diabetic skin lesions through different treatment methods such as hypoglycemic drugs and probiotic emulsions.

Researchers will conduct telephone follow-ups of diabetic patients, collect data, and statistically analyze the impact of changes in the skin microecology of diabetic patients on the occurrence of diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Surface skin cotton swab collection

(1) Observation group: In the endocrinology department of Nanfang hospital, the patient were diagnosed with type 2 diabetes to the WHO 1999 diagnostic criteria for diabetes.

(2) Control group:

1. Control subjects that was ruled out diabetes according to the WHO 1999 diagnostic criteria for euglycemia.
2. Age ≥18 years, the patient and (or) his family members know and agree to participate in this study.

2. Skin tissue collection

(1) Observation group:

1. The patient was diagnosed with type 2 diabetes in the Endocrinology Department, Burns Department, Traumatology Orthopedics, Plastic Surgery in Nanfang hospital.
2. Patients who need surgical operations such as debridement and amputation below the knee joint due to various reasons such as diabetic foot osteomyelitis, fractures, car accidents and so on.

(2) Control group:

1. The patient without type 2 diabetes in the Endocrinology Department, Burns Department, Traumatology Orthopedics, Plastic Surgery in Nanfang hospital.
2. Patients who need surgical operations such as debridement and amputation below the knee joint due to various reasons such as post-traumatic foot osteomyelitis, fractures, car accidents and so on.
3. Age ≥18 years, the patient and (or) his family members know and agree to participate in this study.

Exclusion Criteria:

The patients Including other skin diseases, using medically prescribed soap for bathing, using cosmetics on the feet, suffering from severe liver and kidney disease, immune system disease, HIV infection, malignant tumors, or using immunosuppressive drugs within the first four weeks. The patient or (and) their family members refused to participate in this study.

The researchers judged that they are not suitable to participate in this research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 cases, 40 cases in each group
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
omics analysis of skin microbiome | from September 2020 to July 2021
  Compared with non-diabetic patients, the differences in skin microbiome of diabetic patients with different disease progression.
change of skin pathology in DM | From August 2021 to July 2024
  The pathological changes of the skin tissues of diabetic patients with different disease progression.
The incidence of developing into diabetic foot among the groups | From August 2023 to July 2025
  Follow-up for 2 years to assess the impact of changes in the skin microecology of diabetic patients on the occurrence of diabetic foot ulcers

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi C, Luo X, Huang J, Kong D, Zhang Y, Zou M, Zhou H. Prevalence of S. aureus and/or MRSA in hospitalized patients with diabetic foot and establishment of LAMP methods for rapid detection of the SCCmec gene. BMC Microbiol. 2024 Jan 26;24(1):36. doi: 10.1186/s12866-024-03196-6. PMID 38279164
- [Derived] Zhang S, Li S, Huang J, Ding X, Qiu Y, Luo X, Meng J, Hu Y, Zhou H, Fan H, Cao Y, Gao F, Xue Y, Zou M. Gram-Negative Bacteria and Lipopolysaccharides as Risk Factors for the Occurrence of Diabetic Foot. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2604-2614. doi: 10.1210/clinem/dgad178. PMID 36974462